CLINICAL TRIAL: NCT01712815
Title: Development of an In Vivo Cell Proliferation Marker for PET Assessment of Chemotherapeutic Response in Cancer
Brief Title: PET/CT in Evaluating Response to Chemotherapy in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1B-11-9; NCI-2012-02041 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: HER2-positive Breast Cancer; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (fluorine F 18-clevudine PET/CT) (Experimental): Patients receive fluorine F18-clevudine IV over 1 minute and then undergo PET/CT scan at baseline. Patients with HER2+ breast cancer also undergo fluorine F 18-clevudine PET/CT scan 2-3 weeks after the first course of treatment and after completion of treatment.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Other: questionnaire administration; Radiation: fluorine F 18-clevudine; Procedure: positron emission tomography/computed tomography

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: questionnaire administration — Ancillary studies
Radiation: fluorine F 18-clevudine — Undergo fluorine F 18-clevudine PET/CT scan
  Other Names: 18F-2'-fluoro-5-methyl-1-beta-D-arabinofuranosyluracil-clevudine; 18F-FMAU
Procedure: positron emission tomography/computed tomography — Undergo fluorine F18-clevudine PET/CT scan

SUMMARY:
This phase I trial studies the side effects of positron emission tomography (PET)/computed tomography (CT) in evaluating response to chemotherapy in patients with breast cancer. Comparing results of diagnostic procedures done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Study fludeoxyglucose [18F] 2'-fluoro-5-methyl-1-beta-D-arabinofuranosyluracil-clevudine (FMAU) (fluorine F 18-clevudine ) in 10 patients with known breast cancer to obtain data on safety, circulating metabolite, tumor imaging feasibility, and radiation dosimetry. II. Assess the potential utility of FMAU-PET in the imaging evaluation of chemotherapeutic response in 15 patients with breast cancer. OUTLINE: Patients receive fluorine F18-clevudine intravenously (IV) over 1 minute and then undergo PET/CT scan at baseline. Patients with human epidermal growth factor receptor 2 positive (HER2+) breast cancer also undergo fluorine F 18-clevudine PET/CT scan 2-3 weeks after the first course of treatment and after completion of treatment. After completion of study treatment, patients are followed up at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for Aim 1:
* Scheduled to receive therapy with trastuzumab plus chemotherapy as part of standard care
* Have one or more breast tumors visualized by conventional PET/CT, CT or magnetic resonance imaging (MRI) prior to the PET FMAU study; PET/CT should be within a week prior to 18-F FMAU

Inclusion criteria for Aim 2:

* Have been diagnosed with a HER2+ invasive cancer of the breast
* Scheduled to receive pre-operative therapy with trastuzumab plus chemotherapy as part of standard care
* Have one or more breast tumors visualized by conventional PET/CT, CT or MRI prior to the PET FMAU study; PET/CT should be within a week prior to 18-F FMAU

Exclusion Criteria:

* Have undergone chemotherapy or radiation therapy within the previous one month
* Women of childbearing potential, unless they have had a negative urine human chorionic gonadotropin (HCG) within the previous 24 hours of the procedure
* Patients who have had surgery at the site of the suspected lesion within 1 month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change of FMAU-PET score vs. change of Ki-67 from the baseline to post-chemotherapy | Up to 1 year
Incidence of adverse events | Up to 24 hours after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Conti, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States